CLINICAL TRIAL: NCT05712161
Title: Use of DurAVR™ THV System in Subjects With Severe Aortic Stenosis: Early Feasibility Study
Acronym: DurAVR™ EFS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anteris Technologies Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: SP0028
Record Dates: First submitted 2023-01-13; First posted 2023-02-03 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Aortic Stenosis; Symptomatic Aortic Stenosis; Severe Aortic Valve Stenosis; Aortic Valve Calcification
Keywords: TAVI; TAVR; Transcatheter Valve; Transcatheter Aortic Valve Implantation
MeSH Terms: conditions — Aortic Valve Stenosis; Aortic Valve, Calcification of

STUDY DESIGN:
Intervention Model Description: A prospective, non-randomized, single-arm, multi-center study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- DurAVR™ THV System (Experimental): TAVR procedure
  Interventions: Device: DurAVRTM THV System

INTERVENTIONS:
Device: DurAVRTM THV System — The DurAVR™ Transcatheter Heart Valve (THV) is a balloon expandable transcatheter aortic valve

SUMMARY:
To evaluate the safety and feasibility of DurAVR™ THV System in the treatment of subjects with symptomatic severe native aortic stenosis.

DETAILED DESCRIPTION:
The primary objective is to assess the acute and long-term safety and feasibility of the DurAVR™ device in adult subjects with symptomatic, severe native aortic stenosis eligible for the transcatheter aortic valve replacement as assessed by the Heart Team at the enrolling institutions.

This is a prospective, non-randomized, single-arm, multi-center Study. Subjects will be consented for follow-up to 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are eligible for entry in this study if ALL the following conditions are met:

  1. Symptomatic, severe native aortic stenosis in subjects 65 years or older
  2. Requires aortic valve replacement and is indicated for TAVR as determined by the Heart Team (composed of an experienced interventional cardiologist and an experienced cardiac surgeon)
  3. Eligible for transfemoral delivery of the DurAVR™ THV
  4. Anatomy appropriate to accommodate safe placement of DurAVR™ THV (Preprocedural measurements by TTE and CT required: aortic annulus diameter 21-23 mm by CT)
  5. Understands the study requirements and the treatment procedures and provides written informed consent
  6. Subject agrees to complete all required scheduled follow-up visits.

Exclusion Criteria:

* Subjects are eligible for entry in this study if NONE of the following conditions are met:

Anatomical

1. Anatomy precluding safe placement of DurAVR™ THV
2. Pre-existing prosthetic heart valve in any position
3. Unicuspid or bicuspid aortic valve
4. Severe aortic regurgitation
5. Severe mitral or severe tricuspid regurgitation requiring intervention.
6. Moderate to severe mitral stenosis.
7. Hypertrophic obstructive cardiomyopathy
8. Echocardiographic evidence of intracardiac mass, thrombus or vegetation requiring treatment.
9. Severe basal septal hypertrophy with outflow gradient

   Clinical
10. Evidence of an acute myocardial infarction ≤ 30 days before the intended treatment.
11. Determined inoperable/ineligible for surgery by the Heart Team
12. Any percutaneous coronary or peripheral interventional procedure performed within 30 days prior to the index procedure
13. Blood dyscrasias as defined: leukopenia (WBC < 1000 mm3), thrombocytopenia (platelet count < 50,000 cells/mm3), history of bleeding diathesis or coagulopathy, or hypercoagulable states
14. Untreated clinically significant Coronary Artery Disease (CAD) requiring revascularization
15. Cardiogenic shock manifested by low cardiac output, vasopressor dependence, or mechanical hemodynamic support
16. Need for emergency surgery for any reason
17. Ventricular dysfunction with left ventricular ejection fraction (LVEF) < 30% as measured by resting echocardiogram
18. Recent (within 6 months) cerebrovascular accident (CVA) or transient ischemic attack (TIA).
19. Symptomatic carotid or vertebral artery disease
20. End stage renal disease requiring chronic dialysis or creatinine clearance < 20 cc/min.
21. GI bleeding within the past 3 months
22. A known hypersensitivity or contraindication to any of the following which cannot be adequately pre-medicated: aspirin, heparin, nitinol (titanium or nickel), ticlopidine and clopidogrel, contrast media
23. Ongoing sepsis, including active endocarditis (Duke Criteria) [49]
24. Subject refuses a blood transfusion
25. Life expectancy < 12 months due to associated non-cardiac co-morbid conditions
26. Other medical, social, or psychological conditions that in the opinion of an Investigator precludes the subject from appropriate consent
27. Severe dementia (resulting in either inability to provide informed consent for the trial/procedure, prevents independent lifestyle outside of a chronic care facility, or will fundamentally complicate rehabilitation from the procedure or compliance with follow-up visits)
28. Currently participating in an investigational drug or another investigational device trial
29. Subject is contraindicated for MDCT or MRI Scans.
30. Subject belongs to a vulnerable population (Vulnerable subject populations are defined as individuals with mental disability, persons in nursing homes, children, impoverished persons, homeless persons, nomads, refugees, and those permanently incapable of giving informed consent. Vulnerable populations also may include members of a group with a hierarchical structure such as university students, subordinate hospital and laboratory personnel, employees of the Sponsor, members of the armed forces, and persons kept in detention).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-08-07 (Actual); Primary Completion 2023-12-29 (Actual); Study Completion 2033-12 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality or disabling stroke | 30days
  Mortality would be reported as rate of death/mortality at 30 days. Disabling stroke would be reported according to VARC-3 Guidelines
Technical success | Immediate post procedure
  Freedom from mortality, successful device implant, and freedom from surgery or intervention related to the device.

SECONDARY OUTCOMES:
All-cause mortality | 30days
  Mortality would be reported as rate of death/mortality at 30days.
Disabling stroke | 30days
  Rate of disabling stroke according to VARC-3 Guidelines
Major vascular, access-related, or cardiac structural complication | 30days
  complications according to VARC-3 Guidelines
VARC-3 Type 2-4 bleeding | 30days
  Rates of Type 2, 3, and 4 bleeding according to VARC-3 guidelines
Acute Kidney Injury stage 3 or 4 | 30days
  AKI stage 3-4 according to VARC-3 guidelines
Moderate or severe aortic regurgitation | 30days
  aortic regurgitation according to VARC-3 guidelines
New permanent pacemaker due to procedure related conduction abnormalities | 30days
  Rate of pacemaker interventions in subjects experiencing conduction abnormalities
Surgery or intervention related to the device, including aortic valve reintervention. | 30days
  Device related interventions

OTHER OUTCOMES:
Hospitalization (or re-hospitalization) | 1 year
  Hospitalization (or re-hospitalization). Any admission after the index hospitalization or study enrolment to an inpatient unit or hospital ward for ≥24 h, including an emergency department stay. Hospitalizations planned for pre-existing conditions are excluded unless there is worsening of the baseline condition.
Leaflet thickening and reduced motion | 1year
  Assessing causes of valve leaflet thickening and reduced leaflet motion such as leaflet thrombosis, endocarditis, leaflet deterioration, and valve frame expansion issues.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Reardon, MD, Study Chair — Methodist DeBakey Hospital
Locations (5):
- United States (5):
  - Tucson Medical Center, Tucson, Arizona
  - University of Michigan, Ann Arbor, Michigan
  - Columbia University Medical Center/NYPH, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No